CLINICAL TRIAL: NCT03623958
Title: Image Guided VATS Resection vs. VATS Resection of Lung Lesions
Brief Title: Image Guided VATS vs. VATS Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raphael Bueno, Chief of Throacic Surgery, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000291
Record Dates: First submitted 2018-07-20; First posted 2018-08-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: image guided; lung nodule; lung cancer; lung mass
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iVATS resection (Experimental): Image guided Video-assisted thoracoscopic surgery (VATS) in either one of two hybrid operating rooms and Fine Needle Aspiration (FNA) under fluoroscopy.
  Interventions: Device: Image guided Video-Assisted Thoracic Surgery (VATS) resection
- Standard VATS resection (Active Comparator): Standard video-assisted thoracoscopic surgery (VATS) in operating room and Fine Needle Aspiration (FNA) in pathology frozen section room.
  Interventions: Procedure: Video-Assisted Thoracic Surgery

INTERVENTIONS:
Device: Image guided Video-Assisted Thoracic Surgery (VATS) resection — Image guided placement of a fiducial consisting of a needle directed placement of a T-Bar next to the target lesion in order to lead the surgeon to the lung region to be removed
  Arms: iVATS resection
Procedure: Video-Assisted Thoracic Surgery — Standard of Care Video-Assisted Thoracic Surgery (VATS) resection
  Arms: Standard VATS resection

SUMMARY:
To evaluate workflow and outcomes of iVATS and standard VATS for small pulmonary nodules. The outcomes of the patients will be evaluated separately as there will be no direct comparison of the two arms.

DETAILED DESCRIPTION:
This is a prospective phase II clinical study to evaluate iVATS and standard VATS for small pulmonary nodules. We have successfully completed and published a phase I/pilot study with 25 patients demonstrating safety and optimal procedural workflow for combining image-guidance with VATS. This phase II clinical study will further expand upon the safety and feasibility of this procedure. Additionally, this data will be used to design a phase III comparison study between iVATS and standard VATS.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years and older
* Subject must be deemed a candidate for the iVATS surgery, by their treating Thoracic Surgeon
* Subject must have nodules/GGO or other abnormal opacity that can be accurately measured in at least one dimension with longest diameter ≤ 20 mm or 2cm
* Subject's lesions that are located in the outer half portion of the lung/lobe.
* Subjects must be evaluated at BWH and/or DFCI Thoracic Surgery outpatient clinics

Exclusion Criteria:

* If participant is a pregnant woman or breast feeding they will not be eligible.
* If treating thoracic surgeon deems the participant not eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Operating Room Time | 3 years to complete
  The time (in min.) from incision to close

SECONDARY OUTCOMES:
Time to T-bar placement | 3 years
  The time from patient ready for surgery to placement of t-bar
Time for induction to incision | 3 years
  Time (in min) from induction to incision made
Hospital Length of Stay | 3 years
  Length of hospital stay (in days) in both arms
Radiation Exposure | 3 years
  The radiation exposure (mSV) in the iVATS arm

OTHER OUTCOMES:
Quantitative Analysis of CT scans | 3 years
  To collect imaging data from pre-operative and post-operative CT scans for quantitative analysis from both arm.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Bueno, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Gill RR, Zheng Y, Barlow JS, Jayender J, Girard EE, Hartigan PM, Chirieac LR, Belle-King CJ, Murray K, Sears C, Wee JO, Jaklitsch MT, Colson YL, Bueno R. Image-guided video assisted thoracoscopic surgery (iVATS) - phase I-II clinical trial. J Surg Oncol. 2015 Jul;112(1):18-25. doi: 10.1002/jso.23941. Epub 2015 May 28. PMID 26031893